CLINICAL TRIAL: NCT03268772
Title: Pegylated-liposome Doxorubicin Combined With Ifosfamide As First-line Treatment for Patients With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: PLD and IFO As First-line Treatment for Patients With Advanced or Metastatic STS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Vice professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-STS-01
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLD-IFO (Experimental): pegylated liposomal doxorubicin (PLD) combined with ifosfamide (IFO)
  Interventions: Drug: PLD and IFO

INTERVENTIONS:
Drug: PLD and IFO — PLD 30 mg/m2, d1, plus IFO 1.8 g/m2, d1-5

SUMMARY:
This study is designed to evaluate the efficacy and safety of pegylated liposomal doxorubicin (PLD) combined with ifosfamide (IFO) for the first-line treatment of patients with advanced or metastatic soft tissue sarcoma (STS).

DETAILED DESCRIPTION:
This phase II study is designed to evaluate the efficacy and safety of pegylated liposomal doxorubicin (PLD) combined with ifosfamide (IFO) for the first-line treatment of patients with advanced or metastatic soft tissue sarcoma (STS).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years with histologically confirmed advanced or metastatic STS
* Eastern Cooperative Oncology Group performance status of 0 to 2
* life expectancy of ≥ 3 months
* have not received chemotherapy before
* at least one measurable lesion
* LVEF≥50%
* have adequate bone marrow, hepatic, and renal function

Exclusion Criteria:

* osteosarcoma, Ewing's sarcoma/PNET (primitive neurotodermal tumour),GIST(Gastrointestinal Stromal Tumors), rhabdomyosarcoma, dermatofibrosarcoma protuberans
* patients with symptomatic brain metastases
* active clinical severe infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 6 months

SECONDARY OUTCOMES:
overall response rate | 2 months
overall survival | 12 months
Adverse Events | 2 months
biomarker analysis | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu X, Jiang S, Wang H, Wu X, Yan W, Chen Y, Xu Y, Wang C, Yao W, Wang J, Yu L, Miao J, Chen H, Xia J, Huang M, Zhang X, Luo Z. Pegylated Liposomal Doxorubicin Combined with Ifosfamide for Treating Advanced or Metastatic Soft-tissue Sarcoma: A Prospective, Single-arm Phase II Study. Clin Cancer Res. 2022 Dec 15;28(24):5280-5289. doi: 10.1158/1078-0432.CCR-22-1785. PMID 36239473